CLINICAL TRIAL: NCT02308683
Title: The Effects of Moringa Oleifera Supplements on hsCRP and HgbA1c Levels of Patients in Ospital ng Maynila Medical Center Diabetic Clinic: A Prospective Cohort Study
Brief Title: Effects of Moringa Oleifera on hsCRP and Hgba1c Level of Patients in Ospital ng Maynila Medical Center Diabetic Clinic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ospital ng Maynila Medical Center (Other)
Responsible Party: Principal Investigator, Rainier N. Mozo, The Effects of Moringa oleifera supplements on hsCRP and HgbA1c Levels of Patients in Ospital ng Maynila Medical Center Diabetic Clinic: A Prospective Cohort Study, Ospital ng Maynila Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Moringa oleifera
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes
Keywords: hscrp; hgba1c; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — flocculant protein MO 2.1, Moringa oleifera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hsCRP, Hgba1c (Experimental): Pre treatment hsCRP and hgba1c will be initially measured After 12 weeks supplementation of Moringa oleifera, post treatment hsCRP and Hgba1c will be measured
  Interventions: Dietary Supplement: Moringa oleifera

INTERVENTIONS:
Dietary Supplement: Moringa oleifera — 12 weeks supplementation
  Other Names: Malungay

SUMMARY:
Current evidence supports a central role of inflammation in the pathogenesis of atherosclerosis and diabetes [57-60]. Diabetes Mellitus type 2 is an inflammatory atherothrombotic condition associated with high prevalence of thrombotic cardiovascular disease. In patient with DM type 2, this inflammation is reflected by elevated plasma levels of several biomarkers of inflammation such as C-reactive protein (CRP) [51-55]. HsCRP is considered as a strong predictive of cardiovascular risks and death [53, 61-72]. Besides its predictive role in determining cardiovascular risk, there is some evidence that CRP may represent an active participant in atherogenesis [54]. CRP is expressed in human atherosclerotic plaques and both vascular cells and monocytes/macrophages appear to represent a significant source of CRP in the inflammatory vessel wall [54].

Among the DM risk factors (like hypertension, atherogenic dyslipidemia, insulin resistance, impaired fibrinolysis, inflammatory profile), definitely, inflammation is the neglected one.

Moringa oleifera has been suggested to exert anti-inflammatory effects [42][43][45] and hypoglycemic property [80]. As with many reports of the nutritional or medicinal value of a natural product, there are an alarming number of purveyors of "healthful" food who are now promoting M. oleifera as a panacea. While much of this recent enthusiasm indeed appears to be justified, it is critical to separate scientific evidence from anecdote.

Herein, the investigators will investigate the effects of Moringa oleifera leaves supplementation on levels of inflammatory marker specifically hsCRP, hgbA1c level and clinical outocome in diabetic patients through a cohort study.

DETAILED DESCRIPTION:
We performed a prospective cohort study of adult diabetics who were given 12-weeks supplementation of Moringa oleifera. Plasma hsCRP and serum HgbA1c were compared before and after treatment with M. oleifera.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged between 19 and 65 years of age.
2. They were diagnosed by the Internal Medicine resident or other physician as having Diabetes Mellitus using the following criteria stated by American Diabetes Association (ADA)
3. Participants should be willing to have their blood extracted for hsCRP and Hgba1c measurement before and after 12 weeks supplementation of M. oleifera.
4. Participants have available treatment partner.
5. Subjects who have been diagnosed with other diseases such as asthma, stroke, or hypertension was included in the trial provided since they are already medically stable and that these diseases are not listed as part of the exclusion criteria.

Exclusion Criteria:

1. Subjects who are suspected to have psychiatric disorders, mentally challenged, or confirmed to be pregnant
2. Subjects who are not medically stable or those confirmed to be afflicted with communicable or life threatening diseases such as but not limited to the following:

   * ongoing infection (Pulmonary Tuberculosis, DM foot infection, cellulitis, pneumonia, Urinary Tract Infections, ear infections or dental/gum Infections)
   * decompensated heart failure ( CHF III-IV)
   * chronic liver disease in decompensated state
   * stroke in evolution,
   * acute coronary syndrome within 6 months,
   * systemic or pulmonary inflammatory condition (including rheumatoid arthritis, systemic lupus erythematosus,
   * chronic obstructive pulmonary disease in exacerbation,
   * bronchial asthma in exacerbation, history of renal or other organ transplant and/or
   * immunocompromised state
3. Subjects with anemia (hemoglobin value of less than 13.0 g/dl in males; 12.0 g/dl in females)
4. Subjects with undergoing Moringa oleifera, fish oil or any vitamins or multivitamins supplementation within the past 8 weeks are excluded in the study.
5. Subjects with the use of estrogen/progesterone hormone. Subjects with plan or anticipated by their physicians to be initiated with renal replacement therapy (dialysis) during the study.
6. Subjects who are pregnant or plan to be pregnant.
7. Subjects with known or suspected allergy to M. oleifera or any other component to the drug preparation.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Post treatment mean HsCRP | 12 weeks

SECONDARY OUTCOMES:
Post treatment mean hgba1c | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rainier Mozo, Dr, Principal Investigator — Ospital ng Maynila Medical Center Department of Internal Medicine and ICU